CLINICAL TRIAL: NCT00646516
Title: A Rand, Doubleblind, Activecontrolled, Parallel-grp,Singledummy, Multicenter,12 wk Study to Assess the Effic.&Safety of Symbicort pMDI 2x160/4.5mcg QD Compared to Symb. pMDI 2x80/4.5mcg QD, Symb. pMDI 2x80/4.5mcg Bid and to Budesonide pMDI 2x160 Mcg QD in Asthmatic Sub's12yrs and Over
Brief Title: Gemini Symbicort pMDI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5896C00001
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Mild or Moderate Asthma
Keywords: Asthma; inhaled corticosteroids; Symbicort; budesonide/formoterol; budesonide
MeSH Terms: conditions — Lymphoma, Follicular; Asthma | interventions — Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: budesonide/formoterol (Symbicort)

INTERVENTIONS:
Drug: budesonide/formoterol (Symbicort)
  Other Names: Symbicort

SUMMARY:
The purpose of this study is to determine whether treatment with Symbicort for 12 weeks will improve lung function and symptoms of adults and adolescents with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma
* Baseline lung function tests as determined by protocol.
* Required and received treatment with inhaled corticosteroids and/or lung treatments specified in the protocol within timeframe and doses specified in protocol.

Exclusion Criteria:

* Severe asthma
* Has required treatment with any non-inhaled corticosteroid within previous 4 weeks, has sensitivity to drugs specified in the protocol or requires treatment with beta-blockers
* Had cancer within previous 5 years or currently has any other significant disease or disorder as judged by the investigator

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 615 (Estimated)
Dates: Start 2003-10; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Change from start of treatment in evening pre-dose FEV1 | 2, 6 and 12 weeks after starting treatment

SECONDARY OUTCOMES:
Change from before treatment in lung function, symptoms, use of rescue medication and patient-physician reported outcomes | Daily
Investigate safety profile of Symbicort and budesonide | Before and 2, 4, 12 weeks after start of treatment and 1 week after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Liza O'Dowd, MD, Study Director — AstraZeneca; Catherine Bonuccelli, Study Chair — AstraZeneca

REFERENCES:
- [Derived] Kerwin EM, Oppenheimer JJ, LaForce C, Parasuraman B, Miller CJ, O'Dowd L, Goldman M. Efficacy and tolerability of once-daily budesonide/formoterol pressurized metered-dose inhaler in adults and adolescents with asthma previously stable with twice-daily budesonide/ formoterol dosing. Ann Allergy Asthma Immunol. 2009 Jul;103(1):62-72. doi: 10.1016/S1081-1206(10)60145-7. PMID 19663129